CLINICAL TRIAL: NCT06168604
Title: The Pain Identification and Communication Toolkit: A Training Program to Support Family Caregivers of Persons With ADRD
Brief Title: Evaluating the Efficacy of the Pain Identification and Communication Toolkit
Acronym: PICT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 22-08025205; R01AG079932 (NIH)
Record Dates: First submitted 2023-12-01; First posted 2023-12-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Caregiver Burden; Cognitive Impairment; Dementia; Alzheimer Disease; Pain, Chronic
Keywords: Family Caregivers; Informal Caregivers; Dementia; Pain
MeSH Terms: conditions — Caregiver Burden; Cognitive Dysfunction; Dementia; Alzheimer Disease; Chronic Pain; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single blind allocation. The outcomes assessors will be masked to group allocation. Other research personnel (investigator, project manager, interventionist) may become aware of group allocation. Participants will be asked not to disclose to outcomes assessors the group to which they are assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Identification and Communication Toolkit (Experimental): The Pain Identification and Communication Toolkit (PICT) components include: a) training using an observational assessment tool to detect pain in persons with Alzheimer's disease and related dementias (ADRD), b) coaching and feedback by a trained interventionist in effective strategies for communicating with providers about pain, c) future planning for what steps to take when a pain symptom is detected, and d) updating the caregiver's skill set through routine practice and homework exercises. A trained interventionist will deliver the PICT intervention following a manualized protocol to the caregiver participants. Patient participants will not receive any intervention.
  Interventions: Behavioral: Pain Identification and Communication Toolkit
- Attention Control (Sham Comparator): The Attention Control (AC) condition, also known as the Health Promotion Program (HPP), focuses on caregiver health promotion topics, such as nutrition, exercise, and sleep. A trained interventionist will provide education on these topics using scripted material, use active listening and open questioning techniques, and provide the HPP participants with worksheets (e.g., meal plans) to complete between sessions to mirror the homework activities in the PICT condition for the caregiver participants. Patient participants will not receive any intervention.
  Interventions: Behavioral: Health Promotion Program

INTERVENTIONS:
Behavioral: Pain Identification and Communication Toolkit — The Pain Identification and Communication Toolkit (PICT) is a multicomponent (6 module) intervention for family caregivers of persons with Alzheimer's disease and related dementias (ADRD). PICT consists of 4 weekly telephone sessions (30-60 minutes each) delivered by a trained interventionist
  Arms: Pain Identification and Communication Toolkit
Behavioral: Health Promotion Program — The attention control (AC) condition is referred to as the Health Promotion Program (HPP). The HPP will consist of 4 weekly telephone sessions (30-60 minutes each) but focus on caregiver health promotion topics, such as nutrition, exercise, and sleep.
  Arms: Attention Control

SUMMARY:
This study will evaluate the Pain Identification and Communication Toolkit (PICT), a multicomponent intervention for caregivers of people with Alzheimer's disease and related dementias (ADRD). PICT provides training in observational pain assessment and coaching in effective pain communication techniques. It will recruit participants from programs of all-inclusive care for the elderly (PACE) and partnering health care clinics. The investigators hypothesize that PICT will help caregivers to recognize and communicate about pain in their care recipients.

DETAILED DESCRIPTION:
Up to 60% of older persons with Alzheimer's disease and related dementias (ADRD) suffer from bothersome pain and nearly half experience pain-related activity limitations. Despite best-practice guidelines calling for routine pain assessment of persons with ADRD, pain is severely under-detected and poorly managed in this population. A major barrier to the identification and treatment of pain in persons with ADRD is impaired communication. Informal (family) caregivers are well situated to detect pain and facilitate management in persons with ADRD, given their extensive involvement in care activities. However, caregivers receive virtually no guidance or training in these areas. The Pain Identification and Communication Toolkit (PICT) is a multicomponent intervention for ADRD caregivers that provides training in observational pain assessment and coaching in effective pain communication techniques. PICT consists of 4 weekly telephone sessions (30-60 minutes each) delivered by a trained interventionist. This project aims to (1) determine the efficacy of PICT compared with an Attention Control (AC) condition, (2) identify the patient and caregiver factors that may moderate the effects of PICT on study outcomes, and (3) evaluate the mechanisms (theoretically-derived variables) by which PICT affects study outcomes. Participants will be recruited from programs of all-inclusive care for the elderly (PACE) programs and partnering health care clinics. They will complete assessments at 0 (baseline), 1, 3, and 6 months.

ELIGIBILITY:
CAREGIVER PARTICIPANTS

Inclusion Criteria:

1. Age 21 or older
2. Any gender
3. English speaking
4. Cognitively intact (BOMC ≤10)
5. Provides care to a community-dwelling adult with dementia or cognitive impairment who also has a pain diagnosis
6. Care recipient is not enrolled in hospice
7. Visits the care recipient at least weekly
8. Accessible by telephone

Exclusion Criteria:

1. Paid caregiver
2. Age 20 or younger
3. Non-English speaking
4. Cognitively impaired
5. Does not provide care to a person with dementia or cognitive impairment who also has a pain diagnosis
6. Currently enrolled in hospice
7. The patient to whom the caregiver provides assistance is enrolled in hospice
8. Visits care recipient less than weekly
9. Not accessible by telephone.

PATIENT PARTICIPANTS

Inclusion Criteria:

1. Residing in community settings
2. Record of dementia or cognitive impairment
3. Diagnosis of pain
4. Responsive to environment
5. No terminal illness with life expectancy <6 months
6. Not in active cancer treatment

Exclusion Criteria:

1. Lives in a residential facility (such as a nursing home or assisted living)
2. Enrolled in hospice
3. No dementia or cognitive impairment
4. Unresponsive to environment
5. Has terminal illness with life expectancy <6 months
6. Are in active cancer treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in caregiver-reported pain communication | Baseline, 1 month, 3 month, 6 month
  Change in caregiver-reported pain-related communication as measured by ten questions from the Perceived Involvement in Care Scale (PICS). The range of possible scores is 10-50, where higher scores indicate greater caregiver involvement in patient consultation.
Change in pain management discussions with health care providers | Baseline, 1 month, 3 month, 6 month
  Change in pain management discussions as measured by the combined number of phone calls and appointments made to discuss pain management recorded in the patient's medical chart.
Change in concordance between patient and caregiver pain ratings | Baseline, 1 month, 3 month, 6 month
  Change in concordance in patient and caregiver pain ratings as measured by the absolute difference between caregiver and patient pain ratings of the patient's pain on the Iowa Pain Thermometer (IPT). The IPT is scored on a scale of 0-10 where 0 means "no pain" and 10 means "the most intense pain imaginable."
Change in caregiver's ability to recognize pain | Baseline, 1 month, 3 month, 6 month
  Change in caregiver's ability to recognize pain as measured by the absolute difference between the caregiver-reported PAINAD score and correct PAINAD score (i.e. absolute value of the deviance between the scores). The PAINAD is scored on a scale from 0-10 where 0 means "no pain" and 10 means "severe pain." Participants will be shown multiple videos on which to score the PAINAD.
Change in caregiver's ability to recognize pain behaviors | Baseline, 1 month, 3 month, 6 month
  Change in caregiver's ability to recognize pain behaviors as measured by the absolute difference between the number of caregiver-reported behaviors within each of the 5 PAINAD behaviors (i.e., Breathing, Negative Vocalization, Facial Expression, Body Language, Consolability) and correct number of behaviors. Participants will be shown multiple videos on which to score the PAINAD.

SECONDARY OUTCOMES:
Change in patient's behavioral disturbance | Baseline, 1 month, 3 month, 6 month
  Change in patient's behavioral disturbance as measured by 11 items on the Memory and Behavior Problem Checklist. Questions are asked on a likert scale of 0-never occurs to 4-occurs daily or more often for a total possible score of 44, with higher scores indicating more behavioral disturbance in the patient.
Change in patient's pain treatments or regimens | Baseline, 1 month, 3 month, 6 month
  Change in number of each type of caregiver-reported patient treatment/regimens.
Change in caregiver burden | Baseline, 1 month, 3 month, 6 month
  Change in caregiver burden will be assessed by the 7-item version of the Zarit Burden Index (ZBI). Response options for each item range from 0-"never" to 4-"nearly always". The highest possible score is 28 and the lowest possible score is 0; higher scores indicate more caregiver burden.
Change in caregiver distress level | Baseline, 1 month, 3 month, 6 month
  Change in caregiver distress as measured by 11 items on the Memory and Behavior Problem Checklist. Questions are asked on a likert scale of 0-not at all to 4-extremely for a highest possible score of 44 and a lowest possible score of 0, with higher scores indicating more caregiver distress.
Change in caregiver self-efficacy in pain recognition | Baseline, 1 month, 3 month, 6 month
  Change in caregiver self-efficacy in pain recognition as measured by 9 items adapted from The Health Education Impact Questionnaire on a scale of 1-"completely disagree" to 5-"completely agree" with a highest total score of 45 and a lowest total score of 9. Higher total scores indicate higher self-efficacy in pain recognition.
Change in caregiver self-confidence in recognizing pain | Baseline, 1 month, 3 month, 6 month
  Change in self-confidence in recognizing pain as measured by four items adapted from McCabe et al., 2012. Questions are asked on a scale of 1-"not at all confident" to 4-"very confident," with a highest possible score of 16 and a lowest possible score of 4. Higher scores indicate more confidence in ones ability to recognize pain.
Change in caregiver self-efficacy in pain-related communication | Baseline, 1 month, 3 month, 6 month
  Change in caregiver self-efficacy in pain-related communication as measured by a modified 10-item version of the Perceived Efficacy in Patient-Physician Interactions (PEPPI) Scale. Questions are asked on a scale of 1 - "not at all confident" to 5 - "very confident" with a highest total score of 50 and a lowest total score of 10. Higher scores indicate higher self-efficacy in pain-related communication between a caregiver and a healthcare provider.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Riffin, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the study, a complete, cleaned, de-identified copy of the quantitative data components described above (i.e., data from questionnaires and medical chart review) will be incorporated into a computerized, shareable database. This database, along with data dictionaries and data collection forms, will be made available to share with interested external investigators upon completion of the study and by the online publication date of the primary and secondary aims in a peer-reviewed journal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available at the earlier time point: either at time of an associated publication or the end of the grant's performance period. Data will be available for three years following the end of the grant period.
Access Criteria: Data will be shared by the PI in accordance with NIH's data sharing policy. De-identified data will be shared upon request. External investigators will be able to access the data by contacting the PI who will share the curated data. Refined data, after de-identification, will be shared with investigators upon request. External investigators will be able to locate and access the data by contacting the PI who will share the curated dataset (as described above). Datasets from this study will be appropriate for deposit in archives at peer-reviewed journals that require data deposition. The PI agrees to share our data with researchers working under an institution with Federal Wide Assurance who agree to a data sharing agreement that stipulates protection of participant privacy and data confidentiality, that the data will be used for research only, and that data will not be transferred to other users.